CLINICAL TRIAL: NCT04400838
Title: A Phase 2/3 Study to Determine the Efficacy, Safety and Immunogenicity of the Candidate Coronavirus Disease (COVID-19) Vaccine ChAdOx1 nCoV-19
Brief Title: Investigating a Vaccine Against COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: COV002
Record Dates: First submitted 2020-05-12; First posted 2020-05-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Coronavirus
Keywords: Covid-19; ChAdOx1 nCov19; sars-cov-2; vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — ChAdOx1 nCoV-19; Meningococcal Vaccines; Real-Time Polymerase Chain Reaction; PRIME protocol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (29):
- Group 1 a1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs 260)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260)
- Group 1 a3 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine: 5x10^10vp (Abs 260) prime and 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260) boost, minimum 4 weeks from prime
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 1 b1 (Experimental): Volunteers will receive two dose ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs 260) prime and 2.2x10^10vp (qPCR) boost (4-6 weeks apart)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260) + 2.2x10^10vp (qPCR) boost
- Group 2 a1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs 260)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260)
- Group 2 a3 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine: 5x10^10vp (Abs 260) prime and 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260) boost, minimum 4 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 2 b1 (Experimental): .Volunteers will receive two dose ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs 260) prime and 2.2x10^10vp (qPCR) boost 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260) + 2.2x10^10vp (qPCR) boost
- Group 4 a1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCoV19 vaccine, 5x10^10vp (Abs 260)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260)
- Group 4 b1 (Experimental): Volunteers will receive two dose ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs 260) prime and 2.2x10^10vp (qPCR) boost 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260) + 2.2x10^10vp (qPCR) boost
- Group 4 c1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCOV19 vaccine, 5x10^10vp (Abs260) prime and 2.2x10^10vp (qPCR) boost*, at least 4 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 5 a1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCoV19 vaccine, 5x10^10vp, (Abs 260)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260)
- Group 5 a3 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine: 5x10^10vp (Abs 260) prime and 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260) boost, minimum 4 weeks from prime
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 5 b1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCoV19 vaccine, 5x1010vp, (qPCR)
  Interventions: Biological: ChAdOx1 nCoV-19 (qPCR)
- Group 5 c1 (Experimental): Volunteers will receive a single dose ChAdOx1 nCoV19 vaccine, 5x10^10vp, (qPCR)
  Interventions: Biological: ChAdOx1 nCoV-19 (Abs 260)
- Group 5 d1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 5 e1 (Experimental): Two dose ChAdOx1 nCoV-19 0.5mL (Covishield 0.9 x 10^11 vp/mL), 4-6 weeks apart
  Interventions: Biological: Two dose ChAdOx1 nCoV-19/Covishield 0.5mL
- Group 5 f1 (Experimental): Two dose ChAdOx1 nCoV-19 (Covishield 0.9 x 10^11 vp/mL), 0.25mL prime and 0.5mL boost 4-6 weeks apart
  Interventions: Biological: Two dose ChAdOx1 nCoV-19/Covishield 0.25mL & 0.5mL
- Group 6 a1 (Experimental): Volunteers will receive a single dose ofChAdOx1 nCoV19 vaccine, 5x1010vp (qPCR)
  Interventions: Biological: ChAdOx1 nCoV-19 (qPCR)
- Group 6 b1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 5x1010vp (Abs260) prime and 0.5mL (3.5 - 6.5 × 1010 vp, Abs 260)* boost* at least 4 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 7 a1 (Experimental): Volunteers will receive a single dose ChAdOx1nCOV19 vaccine, 5x10^10vp (qPCR)
  Interventions: Biological: ChAdOx1 nCoV-19 (qPCR)
- Group 7 b1 (Experimental): Volunteers will receive two doses of ChAdOx1nCOV19 vaccine, 5x10^10vp (qPCR)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 8 a1 (Experimental): Volunteers will receive a single dose ChAdOx1nCOV19 vaccine, 5x10^10vp (qPCR)
  Interventions: Biological: ChAdOx1 nCoV-19 (qPCR)
- Group 8 b1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 9 a1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 10 a1 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 11 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Group 12 (Experimental): Volunteers will receive two doses of ChAdOx1 nCoV19 vaccine, 0.5mL (3.5 - 6.5 × 10^10 vp, Abs 260)* 4-6 weeks apart
  Interventions: Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost
- Single dose MenACWY (Active Comparator): Groups 1 a2, 2 a2, 4 a2, 5 a2, 5 b2, 5 c2, 6 a2, 7 a2 & 8 a2 will receive a standard single dose of MenACWY vaccine
  Interventions: Biological: MenACWY vaccine
- Two dose MenACWY 4 - 6 weeks (Active Comparator): Groups 1 b2, 2 b2, 4 b2, 5 d2, 7 b2, 8 b2, 9 a2 & 10 a2 will receive two doses of MenACWY 4-6 weeks apart
  Interventions: Biological: Two dose MenACWY vaccine
- Two dose MenACWY minimum 4 weeks (Active Comparator): Groups 1 a4, 2 a4, 4 c2, 5 a4, 6b2 will receive two doses of MenACWY at least 4 weeks apart
  Interventions: Biological: Two dose MenACWY vaccine min. 4 weeks apart

INTERVENTIONS:
Biological: ChAdOx1 nCoV-19 (Abs 260) — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 measured by spectrophotometry at Abs260
  Arms: Group 1 a1; Group 2 a1; Group 4 a1; Group 5 a1; Group 5 c1
Biological: MenACWY vaccine — Standard single dose of MenACWY vaccine
  Other Names: Menveo; Nimenrix
  Arms: Single dose MenACWY
Biological: ChAdOx1 nCoV-19 (Abs 260) + 2.2x10^10vp (qPCR) boost — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 measured by spectrophotometry at Abs260 and 2.2x10^10vp ChAdOx1 nCoV-19 boost measured by qPCR 4-6 weeks later
  Arms: Group 1 b1; Group 2 b1; Group 4 b1
Biological: Two dose MenACWY vaccine — Two standard doses of MenACWY vaccine 4-6 weeks apart
  Other Names: Menveo; Nimenrix
  Arms: Two dose MenACWY 4 - 6 weeks
Biological: ChAdOx1 nCoV-19 (qPCR) — A single dose of 5x10^10vp of ChAdOx1 nCoV-19 measured by qPCR
  Arms: Group 5 b1; Group 6 a1; Group 7 a1; Group 8 a1
Biological: ChAdOx1 nCoV-19 0.5mL prime plus boost — Two dose ChAdOx1 nCoV-19 0.5mL (3.5 - 6.5 × 10^10 vp Abs 260)
  Arms: Group 1 a3; Group 10 a1; Group 11; Group 12; Group 2 a3; Group 4 c1; Group 5 a3; Group 5 d1; Group 6 b1; Group 7 b1; Group 8 b1; Group 9 a1
Biological: Two dose MenACWY vaccine min. 4 weeks apart — Two standard doses of MenACWY vaccine minimum 4 weeks apart
  Other Names: Menveo; Nimenrix
  Arms: Two dose MenACWY minimum 4 weeks
Biological: Two dose ChAdOx1 nCoV-19/Covishield 0.5mL — Two dose ChAdOx1 nCoV-19 0.5mL (Covishield 0.9 x 10^11 vp/mL), 4-6 weeks apart
  Arms: Group 5 e1
Biological: Two dose ChAdOx1 nCoV-19/Covishield 0.25mL & 0.5mL — Two dose ChAdOx1 nCoV-19 (Covishield 0.9 x 10^11 vp/mL), 0.25mL prime and 0.5mL boost 4-6 weeks apart
  Arms: Group 5 f1

SUMMARY:
A phase 2/3 study to determine the efficacy, safety and immunogenicity of the candidate Coronavirus Disease (COVID-19) vaccine ChAdOx1 nCoV-19 in healthy UK volunteers.

DETAILED DESCRIPTION:
There will be 12 study groups and it is anticipated that a total of 12,390 volunteers will be enrolled. Groups 1, 7 & 9 are adults aged 56-69 years; groups 2, 8 & 10 are adults 70 years and over; groups 4, 5 & 6 are adults aged 18-55 years; group 11 is adults aged 18-55 years who have previously received a ChAdOx vectored vaccine; group 12 is HIV positive adults aged 18-55 years.

The vaccine will be administered intramuscularly into the deltoid of the non-dominant arm (preferably).

All subjects will undergo follow-up for a total of 1 year post last vaccination. Additional visits or procedures may be performed at the discretion of the investigators, e.g., further medical history and physical examination, or additional blood tests and other investigations if clinically relevant

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 - 55 years (groups 4, 5, 6 and 11)
* Adults aged 56-69 years (groups 1, 7, and 9)
* Adults aged 70 years and older (groups 2, 8, and 10)
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their General Practitioner and access all medical records when relevant to study procedures.
* For females of childbearing potential only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and vaccination.
* Agreement to refrain from blood donation during the course of the study.
* Provide written informed consent.

Additional Inclusion criteria to Group 12 (HIV sub-study):

* HIV positive
* Receiving antiretroviral therapy
* Undetectable HIV viral load
* CD4>350 cells/mL

Exclusion Criteria:

• Participation in COVID-19 prophylactic drug trials for the duration of the study.

Note: Participation in COVID-19 treatment trials is allowed in the event of hospitalisation due to COVID-19. The COV002 study team should be informed as soon as possible.

• Participation in SARS-CoV-2 serological surveys where participants are informed of their serostatus for the duration of the study.

Note: Disclosure of serostatus post enrolment may accidently unblind participants to group allocation. Participation in COV002 can only be allowed if volunteers are kept blinded to their serology results from local/national serological surveys

* Receipt of any vaccine (licensed or investigational) other than the study intervention within 30 days before and after each study vaccination, with the exception of the licensed seasonal influenza vaccination and the licensed pneumococcal vaccination. Participants will be encouraged to receive these vaccinations at least 7 days before or after their study vaccine.
* Prior or planned receipt of an investigational or licensed vaccine or product likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccines, any coronavirus vaccines). This exclusion criteria will not apply to group 11, as recruitment will be targeted at those volunteers who previously received a ChAdOx1 vectored vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Any confirmed or suspected immunosuppressive or immunodeficient state (except group 12, where HIV infected participants are allowed); asplenia; recurrent severe infections and use of immunosuppressant medication within the past 6 months, except topical steroids or short-term oral steroids (course lasting ≤14 days)
* History of allergic disease or reactions likely to be exacerbated by any component of ChAdOx1 nCoV-19 or MenACWY
* Any history of angioedema.
* Any history of anaphylaxis.
* Pregnancy, lactation or willingness/intention to become pregnant during the study.
* Current diagnosis of or treatment for cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition likely to affect participation in the study.
* Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.
* Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e. warfarin) or novel oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran and edoxaban)
* Suspected or known current alcohol or drug dependency.
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed)
* History of laboratory confirmed COVID-19 (except groups 5d, 5e, 5f, 9, 10 and 11).
* Seropositivity to SARS-CoV-2 before enrolment (except groups 5d, 5e, 5f, 9, 10 and 11)
* NB: volunteers with previous NAAT positive results are also allowed in groups 9, 10 and 11

Additional Exclusion criteria to Groups 4, 6, 9 and 10

* History of allergic disease or reactions likely to be exacerbated by Paracetamol
* Note: Caution should be taken when recommending paracetamol to adults who already take paracetamol chronically

Re-vaccination exclusion criteria (two-dose groups only)

* Anaphylactic reaction following administration of vaccine
* Pregnancy. An exception to this will be prior to receipt of a booster dose at extra visit B. If a pregnant woman has discussed vaccination with their usual clinician (e.g. GP) and chooses to receive a COVID-19 vaccination, this may be administered by the trial team as part of extra visit B. (Protocol 19.0) or as part of the provision of treatment to controls.
* Any AE that in the opinion of the Investigator may affect the safety of the participant or the interpretation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10811 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of the candidate ChAdOx1 nCoV-19 against COVID-19 in adults aged 18 years and older. | Study duration (12 months from last vaccination)
  Number of virologically confirmed (PCR or NAAT positive) symptomatic cases of COVID-19
Assess the safety of the candidate vaccine ChAdOx1 nCoV-19 in adults | Study duration (12 months from last vaccination)
  Occurrence of serious adverse events (SAEs) throughout the study duration.

SECONDARY OUTCOMES:
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV-19: occurrence of solicited local reactogenicity signs and symptoms for 7 days following | 7 days post vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following vaccination
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV-19: occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following | 7 days post vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following vaccination
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV-19: occurrence of unsolicited adverse events (AEs) for 28 days following vaccination | 28 days post vaccination
  Occurrence of unsolicited adverse events (AEs) for 28 days following vaccination
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV-19 through standard blood tests (full blood count, liver and kidney function tests) | 6 months
  Frequency of participants with clinically significant changes from baseline for safety laboratory measures (haematology and biochemistry blood results; except groups 4, 6, 9 & 10)
Assess the safety, tolerability and reactogenicity profile of the candidate vaccine ChAdOx1 nCoV-19 by measuring the number of disease enhancement episodes | Study duration (12 months from last vaccination)
  Occurrence of disease enhancement episodes
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19: hospital admissions | Study duration (12 months from last vaccination)
  Number of hospital admissions associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 | 6 months
  Number of intensive care unit (ICU) admissions associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19: number of deaths | 6 months
  Number of deaths associated with COVID-19
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by measuring seroconversion rates | 6 months
  Proportion of people who become seropositive for non-Spike SARS-CoV-2 antigens during the study
Assess efficacy of the candidate ChAdOx1 nCoV-19 against severe and non-severe COVID-19 by measuring incidence of Covid-19 | Study duration (12 months from last vaccination)
  Proportion of people diagnosed with severe Covid-19 disease (defined according to clinical severity scales)
Assess humoral immunogenicity of ChAdOx1 nCoV-19: antibody quantification | 28 days post vaccination
  Quantify antibodies against SARS-CoV-2 spike protein (seroconversion rates)
Assess humoral immunogenicity of ChAdOx1 nCoV-19: seroconversion | 28 days post vaccination
  Proportion of seroconversion to antibodies against SARS-CoV-2 spike protein at Day 28 post-vaccination
Assess cellular and humoral immunogenicity of ChAdOx1 nCoV-19 through ELISpot assays (groups 1, 2, 7 and 8 only) | 6 months
  Interferon-gamma (IFN-γ) enzyme-linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1, 2, 7 and 8 only): local reactogenicity | 7 days post vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following booster vaccination
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1 and 2 only): systemic reactogenicity | 7 days post vaccination
  Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following booster vaccination
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1 and 2 only) | 28 days post vaccination
  Occurrence of unsolicited adverse events (AEs) for 28 days following booster vaccination
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1 and 2 only) through standard blood tests (full blood count, liver and kidney function tests) | 6 months
  Frequency of participants with clinically significant changes from baseline from pre-booster for safety laboratory measures (haematology and biochemistry blood results)
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1 and 2 only) via seroconversion | 56 days post vaccination
  Antibodies against SARS-CoV-2 spike protein at Day 56 post-vaccination (seroconversion rates)
Assess the safety and immunogenicity of a booster dose of ChAdOx1 nCoV-19 in older adults aged 56 years or older (two-dose schedules for groups 1 and 2 only) | 56 days post vaccination
  Proportion of seroconversion to antibodies against SARS-CoV-2 spike protein at Day 56 post-vaccination

OTHER OUTCOMES:
Exploratory Immunology by virus neutralising antibody assays | 6 months
  Virus neutralising antibody (NAb) assays against live and/or pseudotype SARS-CoV-2 virus
Exploratory Immunology by flow cytometry | 6 months
  Cell analysis by flow cytometry assays
Exploratory Immunology by functional antibody assays | 6 months
  Functional antibody assays
Exploratory Immunology: anti-vector immunity | 6 months
  Anti-vector immunity induced by 1 or 2 doses of ChAdOx1 nCoV-19
Measure exposure to COVID-19 | 6 months
  Reported by weekly survey to collect information about cases amongst household contacts and friends, contact with the general public, infection control procedures
Exploratory efficacy against infection: assess efficacy of the candidate ChAdOx1 nCoV-19 against SARS-CoV-2 infection by PCR or NAAT | 6 months
  Number of PCR or NAAT positive cases of COVID-19 infection
Exploratory efficacy against infection: assess efficacy of the candidate ChAdOx1 nCoV-19 against SARS-CoV-2 infection | 6 months
  Measure of differences in viral loads between those with severe, mild, and asymptomatic PCR+ SARS-CoV-2 infections
Compare safety, reactogenicity and immunogenicity between different manufacturing batches of ChAdOx1 nCoV-19 used in COV001 and COV002 | 6 months
  Differences in safety, reactogenicity and immunogenicity profiles between Group 1 in COV001 and Group 5 in COV002 (proportion of Grade 3 solicited AEs, occurrence of fevers, seroconversion rates at D28, neutralising antibody titres and differences in T-cell responses at D14).
Compare safety, reactogenicity and immunogenicity between different methods for measuring doses | 6 months
  Differences in safety, reactogenicity and immunogenicity profiles between Groups 1, 2, and 5A compared with Groups, 7, 8, and 5B, C and D respectively (proportion of Grade 3 solicited AEs, occurrence of fevers, seroconversion rates at D28, neutralising antibody titres and differences in T-cell responses at D14).
Assess vaccine induced mucosal immunity: Nasal mucosa IgA levels at D0 and D28 in a subset of individuals | 6 months
  Nasal mucosa IgA levels at D0 and D28 in a subset of individuals
Compare viral shedding on stool samples of SARS-CoV-2 PCR or NAAT positive individuals | 6 months
  Differences in viral shedding on stool at 7 days and beyond post SARS-CoV-2 PCR or NAAT positivity
Compare immunogenicity of ChAdOx1 nCoV-19 in participants receiving 1 or 2 doses in groups 1, 2, 7 and 8: differences in antibody titres | 6 months
  Differences in antibody titres (ELISA and Neutralising antibodies) in participants who received 1 or 2 doses of ChAdOx1 nCoV-19 (groups 1, 2, 7 and 8)
Compare immunogenicity of ChAdOx1 nCoV-19 in participants receiving 1 or 2 doses in groups 1, 2, 7 and 8: longevity of immune responses | 6 months
  Longevity of immune responses in participants who received 1 or 2 doses of ChAdOx1 nCoV-19
Describe the impact of previous vaccination with other ChAdOx1 vectored vaccines on safety and immune responses to ChAdOx1 nCoV-19 | 6 months
  Differences reactogenicity profile, antibody titres and T-cell responses between groups 5d and 11 and their relationship with anti-vector neutralising antibody titres.
Assess the cell-mediated and humoral immunogenicity profile of ChAdOx1 nCoV-19 vaccine in HIV infected adults | 6 months
  Cell-mediated and humoral responses against SARS-Cov-2 These will be measured by the following:
  1. Proportion of seroconversion to antibodies (Ab) against SARS-CoV-2 spike protein measured by ELISA.
  2. Interferon-gamma enzyme linked immunospot (ELISpot) responses to SARS-CoV-2 spike protein
  3. Intracellular Cytokine analyses of CD4 and CD8-specific SARS-CoV-2 spike protein responses
  4. Further exploratory immunology including immune responses to a further dose administered via the NHS national roll out
Assess whether increasing age and or CD4 nadir are associated with a lack of immune response in HIV infected adults: CD4 count-vaccine immune responses | 6 months
  Relationship between nadir CD4 count vs vaccine immune responses
Assess whether increasing age and or CD4 nadir are associated with a lack of immune response in HIV infected adults: age vs vaccine immune responses | 6 months
  Relationship between age at enrolment and vaccine immune response
Assess whether increasing age and or CD4 nadir are associated with a lack of immune response in HIV infected adults | 6 months
  Immune responses to ChAdOx1 nCoV-19 (assessed as described above)
Assess the safety of the candidate vaccine ChAdOx1 nCoV-19 in HIV infected adults | Study duration (12 months from last vaccination)
  Measured by the following:
  1. Occurrence of serious adverse events (SAEs) throughout the study duration
  2. Occurrence of solicited local reactogenicity signs and symptoms for 7 days following vaccination
  3. Occurrence of solicited systemic signs and symptoms for 7 days following each vaccination
  4. Occurrence of unsolicited AEs for 28 days following each vaccination
To assess Impact of vaccination on HIV reservoirs | Study duration (12 months from last vaccination)
  Change in Total HIV DNA copies per million CD4 T cells
To assess immunological correlates of protection in relation to occurrence of COVID-19 disease in ChAdOx1 nCoV-19 recipients | Throughout the study, average of 18 months]
  Immunological endpoints (antibody & cellular responses to SARS-COV2 spike protein) and COVID-19 disease endpoints (SARS-COV2 PCR positivity plus symptoms) in ChAdOx1 nCoV-19 recipients

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, Prof, Principal Investigator — University of Oxford
Locations (20):
- United Kingdom (20):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Castle Hill Hospital, Cottingham, Hull
  - St Georges University Hospital NHS Foundation Trust, London, Tooting
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - North Bristol NHS Trust, Bristol
  - NIHR Cambridge Clinical Research Facility, Cambridge
  - NHS Lothian, Western General Hospital, Edinburgh
  - Glasgow University and NHS Greater Glasgow & Clyde, New Lister Building, Glasgow Royal Infirmary & Queen Elizabeth University Hospital, Glasgow
  - Liverpool School of Tropical Medicine (LSTM), Accelerator Research Clinic. Clinical Sciences Accelerator, Liverpool
  - London North West University Healthcare Trust (LNWUH), Northwick Park Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, Department of Infection, St Thomas Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Royal Victoria Infirmary, Newcastle upon Tyne
  - Public Health Wales, Newport
  - University of Nottingham Health Service, Cripps Health Centre, University Park, Nottingham
  - CCVTM, University of Oxford, Churchill Hospital, Oxford
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospitals, Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Ogbe A, Pace M, Bittaye M, Tipoe T, Adele S, Alagaratnam J, Aley PK, Ansari MA, Bara A, Broadhead S, Brown A, Brown H, Cappuccini F, Cinardo P, Dejnirattisai W, Ewer KJ, Fok H, Folegatti PM, Fowler J, Godfrey L, Goodman AL, Jackson B, Jenkin D, Jones M, Longet S, Makinson RA, Marchevsky NG, Mathew M, Mazzella A, Mujadidi YF, Parolini L, Petersen C, Plested E, Pollock KM, Rajeswaran T, Ramasamy MN, Rhead S, Robinson H, Robinson N, Sanders H, Serrano S, Tipton T, Waters A, Zacharopoulou P, Barnes E, Dunachie S, Goulder P, Klenerman P, Screaton GR, Winston A, Hill AV, Gilbert SC, Carroll M, Pollard AJ, Fidler S, Fox J, Lambe T, Frater J. Durability of ChAdOx1 nCoV-19 vaccination in people living with HIV. JCI Insight. 2022 Apr 8;7(7):e157031. doi: 10.1172/jci.insight.157031. PMID 35192543
- [Derived] Flaxman A, Marchevsky NG, Jenkin D, Aboagye J, Aley PK, Angus B, Belij-Rammerstorfer S, Bibi S, Bittaye M, Cappuccini F, Cicconi P, Clutterbuck EA, Davies S, Dejnirattisai W, Dold C, Ewer KJ, Folegatti PM, Fowler J, Hill AVS, Kerridge S, Minassian AM, Mongkolsapaya J, Mujadidi YF, Plested E, Ramasamy MN, Robinson H, Sanders H, Sheehan E, Smith H, Snape MD, Song R, Woods D, Screaton G, Gilbert SC, Voysey M, Pollard AJ, Lambe T; Oxford COVID Vaccine Trial group. Reactogenicity and immunogenicity after a late second dose or a third dose of ChAdOx1 nCoV-19 in the UK: a substudy of two randomised controlled trials (COV001 and COV002). Lancet. 2021 Sep 11;398(10304):981-990. doi: 10.1016/S0140-6736(21)01699-8. Epub 2021 Sep 1. PMID 34480858
- [Derived] Frater J, Ewer KJ, Ogbe A, Pace M, Adele S, Adland E, Alagaratnam J, Aley PK, Ali M, Ansari MA, Bara A, Bittaye M, Broadhead S, Brown A, Brown H, Cappuccini F, Cooney E, Dejnirattisai W, Dold C, Fairhead C, Fok H, Folegatti PM, Fowler J, Gibbs C, Goodman AL, Jenkin D, Jones M, Makinson R, Marchevsky NG, Mujadidi YF, Nguyen H, Parolini L, Petersen C, Plested E, Pollock KM, Ramasamy MN, Rhead S, Robinson H, Robinson N, Rongkard P, Ryan F, Serrano S, Tipoe T, Voysey M, Waters A, Zacharopoulou P, Barnes E, Dunachie S, Goulder P, Klenerman P, Screaton GR, Winston A, Hill AVS, Gilbert SC, Pollard AJ, Fidler S, Fox J, Lambe T; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of the ChAdOx1 nCoV-19 (AZD1222) vaccine against SARS-CoV-2 in HIV infection: a single-arm substudy of a phase 2/3 clinical trial. Lancet HIV. 2021 Aug;8(8):e474-e485. doi: 10.1016/S2352-3018(21)00103-X. Epub 2021 Jun 18. PMID 34153264
- [Derived] Emary KRW, Golubchik T, Aley PK, Ariani CV, Angus B, Bibi S, Blane B, Bonsall D, Cicconi P, Charlton S, Clutterbuck EA, Collins AM, Cox T, Darton TC, Dold C, Douglas AD, Duncan CJA, Ewer KJ, Flaxman AL, Faust SN, Ferreira DM, Feng S, Finn A, Folegatti PM, Fuskova M, Galiza E, Goodman AL, Green CM, Green CA, Greenland M, Hallis B, Heath PT, Hay J, Hill HC, Jenkin D, Kerridge S, Lazarus R, Libri V, Lillie PJ, Ludden C, Marchevsky NG, Minassian AM, McGregor AC, Mujadidi YF, Phillips DJ, Plested E, Pollock KM, Robinson H, Smith A, Song R, Snape MD, Sutherland RK, Thomson EC, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Williams CJ, Hill AVS, Lambe T, Gilbert SC, Voysey M, Ramasamy MN, Pollard AJ; COVID-19 Genomics UK consortium; AMPHEUS Project; Oxford COVID-19 Vaccine Trial Group. Efficacy of ChAdOx1 nCoV-19 (AZD1222) vaccine against SARS-CoV-2 variant of concern 202012/01 (B.1.1.7): an exploratory analysis of a randomised controlled trial. Lancet. 2021 Apr 10;397(10282):1351-1362. doi: 10.1016/S0140-6736(21)00628-0. Epub 2021 Mar 30. PMID 33798499
- [Derived] Voysey M, Costa Clemens SA, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Clutterbuck EA, Collins AM, Cutland CL, Darton TC, Dheda K, Dold C, Duncan CJA, Emary KRW, Ewer KJ, Flaxman A, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Galiza E, Goodman AL, Green CM, Green CA, Greenland M, Hill C, Hill HC, Hirsch I, Izu A, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Libri V, Lillie PJ, Marchevsky NG, Marshall RP, Mendes AVA, Milan EP, Minassian AM, McGregor A, Mujadidi YF, Nana A, Padayachee SD, Phillips DJ, Pittella A, Plested E, Pollock KM, Ramasamy MN, Ritchie AJ, Robinson H, Schwarzbold AV, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, White T, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Single-dose administration and the influence of the timing of the booster dose on immunogenicity and efficacy of ChAdOx1 nCoV-19 (AZD1222) vaccine: a pooled analysis of four randomised trials. Lancet. 2021 Mar 6;397(10277):881-891. doi: 10.1016/S0140-6736(21)00432-3. Epub 2021 Feb 19. PMID 33617777
- [Derived] Ewer KJ, Barrett JR, Belij-Rammerstorfer S, Sharpe H, Makinson R, Morter R, Flaxman A, Wright D, Bellamy D, Bittaye M, Dold C, Provine NM, Aboagye J, Fowler J, Silk SE, Alderson J, Aley PK, Angus B, Berrie E, Bibi S, Cicconi P, Clutterbuck EA, Chelysheva I, Folegatti PM, Fuskova M, Green CM, Jenkin D, Kerridge S, Lawrie A, Minassian AM, Moore M, Mujadidi Y, Plested E, Poulton I, Ramasamy MN, Robinson H, Song R, Snape MD, Tarrant R, Voysey M, Watson MEE, Douglas AD, Hill AVS, Gilbert SC, Pollard AJ, Lambe T; Oxford COVID Vaccine Trial Group. T cell and antibody responses induced by a single dose of ChAdOx1 nCoV-19 (AZD1222) vaccine in a phase 1/2 clinical trial. Nat Med. 2021 Feb;27(2):270-278. doi: 10.1038/s41591-020-01194-5. Epub 2020 Dec 17. PMID 33335323
- [Derived] Voysey M, Clemens SAC, Madhi SA, Weckx LY, Folegatti PM, Aley PK, Angus B, Baillie VL, Barnabas SL, Bhorat QE, Bibi S, Briner C, Cicconi P, Collins AM, Colin-Jones R, Cutland CL, Darton TC, Dheda K, Duncan CJA, Emary KRW, Ewer KJ, Fairlie L, Faust SN, Feng S, Ferreira DM, Finn A, Goodman AL, Green CM, Green CA, Heath PT, Hill C, Hill H, Hirsch I, Hodgson SHC, Izu A, Jackson S, Jenkin D, Joe CCD, Kerridge S, Koen A, Kwatra G, Lazarus R, Lawrie AM, Lelliott A, Libri V, Lillie PJ, Mallory R, Mendes AVA, Milan EP, Minassian AM, McGregor A, Morrison H, Mujadidi YF, Nana A, O'Reilly PJ, Padayachee SD, Pittella A, Plested E, Pollock KM, Ramasamy MN, Rhead S, Schwarzbold AV, Singh N, Smith A, Song R, Snape MD, Sprinz E, Sutherland RK, Tarrant R, Thomson EC, Torok ME, Toshner M, Turner DPJ, Vekemans J, Villafana TL, Watson MEE, Williams CJ, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and efficacy of the ChAdOx1 nCoV-19 vaccine (AZD1222) against SARS-CoV-2: an interim analysis of four randomised controlled trials in Brazil, South Africa, and the UK. Lancet. 2021 Jan 9;397(10269):99-111. doi: 10.1016/S0140-6736(20)32661-1. Epub 2020 Dec 8. PMID 33306989
- [Derived] Ramasamy MN, Minassian AM, Ewer KJ, Flaxman AL, Folegatti PM, Owens DR, Voysey M, Aley PK, Angus B, Babbage G, Belij-Rammerstorfer S, Berry L, Bibi S, Bittaye M, Cathie K, Chappell H, Charlton S, Cicconi P, Clutterbuck EA, Colin-Jones R, Dold C, Emary KRW, Fedosyuk S, Fuskova M, Gbesemete D, Green C, Hallis B, Hou MM, Jenkin D, Joe CCD, Kelly EJ, Kerridge S, Lawrie AM, Lelliott A, Lwin MN, Makinson R, Marchevsky NG, Mujadidi Y, Munro APS, Pacurar M, Plested E, Rand J, Rawlinson T, Rhead S, Robinson H, Ritchie AJ, Ross-Russell AL, Saich S, Singh N, Smith CC, Snape MD, Song R, Tarrant R, Themistocleous Y, Thomas KM, Villafana TL, Warren SC, Watson MEE, Douglas AD, Hill AVS, Lambe T, Gilbert SC, Faust SN, Pollard AJ; Oxford COVID Vaccine Trial Group. Safety and immunogenicity of ChAdOx1 nCoV-19 vaccine administered in a prime-boost regimen in young and old adults (COV002): a single-blind, randomised, controlled, phase 2/3 trial. Lancet. 2021 Dec 19;396(10267):1979-1993. doi: 10.1016/S0140-6736(20)32466-1. Epub 2020 Nov 19. PMID 33220855